CLINICAL TRIAL: NCT01200498
Title: A Phase 2, Prospective, Open-Label Study to Determine the Safety and Efficacy of SB939, A Histone Deacetylase Inhibitor, in Subjects With Primary, Post-Polycythemia Vera, or Post-Essential Thrombocythemia Myelofibrosis (PMF; Post-Polycythemia Vera (PV) Myelofibrosis (MF), Or Post- Essential Thrombosis (ET) MF
Brief Title: Study of SB939 in Subjects With Myelofibrosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: S*BIO (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2010-0319
Record Dates: First submitted 2010-09-09; First posted 2010-09-13 (Estimated); Results first posted 2014-01-30 (Estimated); Last update posted 2014-01-30 (Estimated); Status verified 2013-12

CONDITIONS: Myeloproliferative Disorders
Keywords: Primary Polycythemia Vera; Post Polycythemia Vera; Post Essential Thrombocythemia Myelofibrosis; SB939; PMF; post-PV MF; post-ET MF
MeSH Terms: conditions — Myeloproliferative Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- SB939 (Experimental): SB939 starting dose 60 mg by mouth every other day, three times weekly for 3 weeks.
  Interventions: Drug: SB939

INTERVENTIONS:
Drug: SB939 — Starting dose 60 mg by mouth every other day, three times weekly for 3 weeks.

SUMMARY:
The goal of this clinical research study is to learn if SB939 can help to control myelofibrosis. The safety of this drug will also be studied.

DETAILED DESCRIPTION:
The Study Drug:

SB939 is designed to change the DNA (genetic material) of cancer cells. This may keep the cells from growing and cause them to die.

This is the first study in which SB939 is given to patients with myelofibrosis.

Study Drug Administration:

If you are found to be eligible to take part in this study, you will take SB939 by mouth 3 times a week for the first 3 weeks of every 4-week cycle. In some cases, the study doctor may decide your dose can be raised sometime after Cycle 1.

SB939 can be taken at any time of day, 2 hours before or 2 hours after a meal. You should take SB939 at about the same time each day. Do not open, break, or chew the capsules.

If you have any side effects, the doctor may change the amount or how often you take SB939.

You will fill out a study drug diary to keep track of your SB939 doses. You should bring the diary and all used and unused bottles of study drug with you to every study visit.

Study Visits:

At every study visit, you will be asked about any side effects you have had and any drugs you may be taking.

On Day 1 of Cycle 1 (+/- 3 days):

* You will have a physical exam, including measurement of your vital signs.
* You will be asked about any blood transfusions you have had and drugs you have taken since the last visit.
* Your performance status will be recorded.
* Blood (about 4 teaspoons) will be drawn for routine tests.
* You will have an ECG before taking this medication, about 10 minutes after taking medication, and 4-6 hours after taking medication.

On Day 8 of Cycle 1 (+1-3 days), blood (about 2 teaspoons) will be drawn for routine tests.

On Day 15 of Cycle 1 (+/- 3 days):

* You will have a physical exam, including measurement of your vital signs.
* Blood (about 4 teaspoons) will be drawn for routine tests.
* You will have an ECG before taking this medication, about 10 minutes after taking medication, and 4-6 hours after taking medication.

On Day 22 of Cycle 1 (+1-3 days), blood (about 2 teaspoons) will be drawn for routine tests.

On Day 1 of Cycles 2 and 3 (+/- 3 days):

* You will have a physical exam, including measurement of your vital signs.
* You will be asked about any blood transfusions you have had since the last visit.
* Your performance status will be recorded.
* Blood (about 4 teaspoons) will be drawn for routine tests.
* You will have an ECG.

On Day 1 of Cycles 4 and beyond (+/- 3 days), or every 3 cycles starting on Day 1 of Cycle 6 (+/- 3 days) if the doctor decides your schedule can change (if you have not had serious side effects):

* You will have a physical exam, including measurement of your vital signs.
* You will be asked about any blood transfusions you have had and drugs you have taken since the last visit.
* Your performance status will be recorded.
* Blood (about 4 teaspoons) will be drawn for routine tests.
* You will have a bone marrow biopsy and aspiration to check the status of the disease, if the doctor thinks it is needed.
* You will have an ECG at every visit to MD Anderson.

If your study visit schedule is changed to every 3 cycles (Day 1 of Cycles 6, 9, and so on), blood (about 4 teaspoons) will be drawn for routine tests every 28 days (+/- 3 days). These tests will be done at your local doctor's office. Every 28 days (+/- 3 days), the study staff will also call you to ask how you are doing and if you have had any side effects.

You may have additional bone marrow biopsies and aspirations and ECGs any time the doctor thinks it is needed. The study visits may also occur more often than described above, if the doctor thinks it is needed.

Length of Study:

You may continue taking the study drug for as long as the doctor thinks it is in your best interest. You will no longer be able to take the study drug if the disease gets worse, if intolerable side effects occur, or if you need radiation therapy, surgery, or other chemotherapy.

Your participation on the study will be over once you have completed the end-of-treatment visit and follow-up.

End-of-Treatment Visit:

After you stop taking the study drug for any reason, the following tests and procedures will be performed:

* You will have a physical exam, including measurement of your vital signs.
* You will be asked about any blood transfusions you have had and drugs you have taken since the last visit.
* Your performance status will be recorded.
* Blood (about 4 teaspoons) will be drawn for routine tests.
* You will have a bone marrow biopsy and aspiration to check the status of the disease, if the doctor thinks it is needed.

Follow-up:

The study staff will call you 30 days and 60 days after your last dose of the study drug (+/- 3 days). You will be asked how you are doing and if you have had any side effects.

If you have any side effects within 60 days after you stop taking the study drug, you may have extra tests and procedures. For example, blood (about 2 teaspoons) may be drawn for routine tests. If you are still having side effects, the study staff will continue calling you to ask how you are doing until the side effects get better. The schedule for how often you are called will depend on the side effects.

This is an investigational study. SB939 is not FDA approved or commercially available. It is currently being used for research purposes only.

Up to 41 patients will take part in this study. All will be enrolled at the University of Texas (UT) MD Anderson Cancer Center.

ELIGIBILITY:
Inclusion Criteria:

1. Must be equal to or greater than 18 years of age
2. Must be diagnosed with Primary Myelofibrosis (PMF) or Post-Essential Thrombocythemia (ET) Myelofibrosis (MF) Post-Polycythemia Vera (PV) MF with intermediate-1, intermediate -2 or high risk disease according to the International Working Group (IWG) prognostic scoring system, or if with low risk disease then with symptomatic splenomegaly that is equal to or greater than 5 cm below left costal margin by physical exam.
3. Must have adequate organ function as demonstrated by the following: • alanine aminotransferase (ALT) (SGOT) and/or aspartate aminotransferase (AST) (SGPT) equal to or less than 2.5 times upper limit of normal (ULN), [unless upon judgment of the treating physician, it is believed to be due to extramedullary hematopoiesis (EMH) related to MF] • Total bilirubin equal to or less than 1.5 times ULN • Serum creatinine equal to or less than 2.5 mg/dL
4. Eastern Cooperative Oncology Group (ECOG) performance status (PS) of 0, 1, or 2
5. At least 2 weeks from prior MF-directed treatment (till the start of study drug)
6. Treatment-related toxicities from prior therapies must have resolved to Grade equal to or less than 1
7. No other active malignancies.
8. Females of childbearing potential (a sexually mature woman who: 1) has not undergone a hysterectomy or bilateral oophorectomy; or 2) has not been naturally postmenopausal for at least 24 consecutive months (i.e., has had menses at any time in the preceding 24 consecutive months)).must have negative pregnancy test.

Exclusion Criteria:

1. Prolongation of the QTc interval to >470 msec at baseline ECG
2. Known positive status for HIV, or known active hepatitis A, B, or C infection.
3. Any serious medical condition or psychiatric illness that would prevent, (as judged by the treating physician) the subject from signing the informed consent form or any condition, including the presence of laboratory abnormalities, which places the subject at unacceptable risk if he/she were to participate in the study or confounds the ability to interpret data from the study.
4. Pregnant or lactating females.
5. Current use of drugs known to prolong QTc interval.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2010-11; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alfonso Quintas-Cardama, MD, Principal Investigator — UT MD Anderson Cancer Center
Locations (1):
- UT MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Result] Quintas-Cardama A, Kantarjian H, Estrov Z, Borthakur G, Cortes J, Verstovsek S. Therapy with the histone deacetylase inhibitor pracinostat for patients with myelofibrosis. Leuk Res. 2012 Sep;36(9):1124-7. doi: 10.1016/j.leukres.2012.03.003. Epub 2012 Apr 2. PMID 22475363
- See also: UT MD Anderson Cancer Center official website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: 11/9/2010 through 11/12/2012. All participants recruited at The University of Texas MD Anderson Cancer Center.
Pre-assignment Details: Of the twenty-three participants enrolled, one participant withdrew consent and was excluded before starting the study.
Period: Overall Study
Arm/Group | SB939
Started | 22
Completed | 22
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- SB939: SB939 starting dose 60 mg by mouth every other day, 3 times weekly for 3 weeks.
Arm/Group | SB939
Number analyzed (Participants) | 22
Age, Continuous [Median (Full Range); unit: years] | 67 [51 to 74]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17
  Male | 5
Region of Enrollment [Number; unit: participants]
  United States | 22

OUTCOME MEASURES:

1. Primary Outcome: Participants With an Objective Response
Description: Objective response defined as Complete, Partial response, and Clinical Improvement based on International Working Group (IWG) Criteria: Complete remission (CR): Absence transfusion & growth factor support AND Complete resolution disease-related symptoms/signs; Peripheral blood count remission; Normal leukocyte differential; Bone marrow histological remission. Partial remission (PR): All CR except bone marrow histological remission. Clinical improvement (CI): No CR/PR, disease progression with one: ≥2 g/dL increase hemoglobin level or transfusion independent; Either ≥50% reduction in palpable splenomegaly of spleen ≥10 cm baseline or spleen palpable at >5 cm baseline becomes not palpable; ≥100% increase in platelet count & absolute platelet count ≥50,000 x 10^9/L; or ≥100% increase in absolute neutrophil count (ANC) & ANC ≥0.5 x 10^9/L. Progressive disease: Progressive splenomegaly or Leukemic transformation confirmed by bone marrow blast of ≥20%; or Increase peripheral blood blast
Time Frame: Baseline to 3 Cycles (84 days)
Measure: Number; unit: Participants
Arm/Group | SB939
Number analyzed (Participants) | 22
Participants
  Complete Response (CR) | 0
  Partial Response (PR) | 0
  Clinical Improvement (CI) | 2

ADVERSE EVENTS:
Time Frame: Adverse events captured from the time of participant consent until 30 days after the last dose of drug. The full study reporting period was two years.
Arm/Group | SB939
Serious Adverse Events (participants affected / at risk) | 1/22
Other Adverse Events (participants affected / at risk) | 20/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SB939 (N=22)
Cognitive Disturbance (Nervous system disorders) | 1 (1)
Muscle Weakness (Nervous system disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SB939 (N=22)
Fatigue (General disorders) | 20 (20)
Peripheral Edema (General disorders) | 4 (4)
Diarrhea (Gastrointestinal disorders) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes